CLINICAL TRIAL: NCT00710190
Title: A Study of Baroreflex Hypertension Therapy in Refractory Hypertension
Brief Title: Device Based Therapy in Hypertension Trial
Acronym: DEBuT-HT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 360004-001
Record Dates: First submitted 2008-07-01; First posted 2008-07-04 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
Keywords: Drug Resistant Hypertension; Refractory Hypertension; High Blood Pressure; Baroreflex Hypertension Therapy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rheos Implant (Experimental)
  Interventions: Device: Rheos Baroreflex Hypertension Therapy System

INTERVENTIONS:
Device: Rheos Baroreflex Hypertension Therapy System — This therapy uses implantable device-based electrical activation of the carotid sinus baroreflex to control blood pressure.

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of the Rheos Baroreflex Hypertension Therapy System in patients with refractory hypertension.

DETAILED DESCRIPTION:
The DEBuT-HT trial will investigate the safety and efficacy of Rheos Baroreflex Hypertension Therapy(TM) in patients with refractory hypertension despite full pharmacologic therapy. Enrolled patients will be carefully assessed prior to receiving a permanently implanted Rheos System. Once the system is implanted, these patients will be followed closely for 1 month to establish baseline information. The Rheos System will be programmed "ON" at the 1 month follow-up and incrementally increased at 2 and 3-month follow-up evaluations. An assessment of safety and efficacy will be made at the 4-month follow-up. Enrolled patients will be followed annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age.
* Have been assessed to have bilateral carotid bifurcations located at or below C3 - C4.
* Have blood pressure greater than or equal to 160 mmHg systolic and/or greater than or equal to 90 mmHg diastolic despite at least two months of full therapy with at least three (3) anti-hypertensive medications, of which at least one (1) must be a diuretic.
* Must be certified by the investigator as compliant to taking full doses of medications.
* Have signed an approved informed consent form for participation in this study.

Exclusion Criteria:

* Have been diagnosed with:

  * Baroreflex failure or significant orthostatic hypotension
  * Cardiac brady arrhythmias or chronic atrial fibrillation
* Have carotid atherosclerosis determined by ultrasound or angiographic evaluation with a stenosis of greater than 50%.
* Have prior surgery or radiation in either carotid sinus region
* Currently have implanted electrical medical devices such as cardiac pacing, defibrillation or neurologic stimulation systems.
* Are pregnant or contemplating pregnancy during the 4-month follow-up period.
* Are on dialysis
* Have hypertension secondary to a treatable cause
* Have clinically significant cardiac valvular disease
* Are unable to comply with protocol requirements.
* Are unlikely to survive the protocol follow-up period
* Are enrolled in another concurrent clinical trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Demonstrate the safety of Rheos(TM) Baroreflex Hypertension Therapy (TM) System by evaluating all adverse events and estimating the system and procedure related adverse event rate. | 4 months post implant
Demonstrate a 10 mmHg decrease from baseline (1-Month office cuff blood pressure) in systolic blood pressure after three months of incrementally optimized therapy. | 4 months post implant

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Baal, PhD, Study Director — CVRx, Inc.
Locations (9):
- University Hospital Hradec Kralove, Hradec Králové, Czechia
- Germany (4):
  - University Hospital Bad Oeynhausen, Bad Oeynhausen
  - Charité Campus Buch, Berlin
  - Uniklinik Essen, Essen
  - University Hospital Hannover, Hanover
- Latvian Centre of Cardiology, Riga, Latvia
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Medical University of Gdansk, Gdansk, Poland
- Inselspital Bern, Bern, Switzerland

REFERENCES:
- See also: Related Info — http://www.cvrx.com